CLINICAL TRIAL: NCT01577251
Title: Registry and Biosample Repository
Brief Title: The Radiation Oncology Registry and Biosample Repository
Status: Recruiting | Type: Observational
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: UPCC 11908
Record Dates: First submitted 2012-04-12; First posted 2012-04-13 (Estimated); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Neoplasia
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma, serum and buffy coat are collected and stored in -80 degree Celsius freezer for future biomarker studies.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this study is to establish a registry and biosample repository (defined as blood, urine, and tumor specimens) in patients with a cancer and/or benign tumor diagnosis undergoing radiotherapy.

ELIGIBILITY:
* Anyone age 18 and above with a cancer and/or benign tumor diagnosis undergoing radiotherapy
* Able to sign consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Anyone age 18 and above with a cancer and/or benign tumor diagnosis undergoing radiotherapy
Sampling Method: Probability Sample
Enrollment: 8000 (Estimated)
Dates: Start 2008-06; Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Health Assessments | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Jay Dorsey, MD, PhD, Principal Investigator — University of Pennsylvania
Locations (4):
- United States (4):
  - Virtua Samson Cancer Center, Moorestown, New Jersey
  - Virtua Health & Wellness Center, Voorhees Township, New Jersey
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania